CLINICAL TRIAL: NCT00500474
Title: Clinical Study of Endolymphatic Sac Drainage With or Without Steroids for Intractable Meniere's Disease
Brief Title: Effects of Endolymphatic Sac Drainage With Steroids for Meniere's Disease
Acronym: EDSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osaka University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tk19661217; tk20090401
Record Dates: First submitted 2007-07-11; First posted 2007-07-12 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Meniere's Disease
Keywords: Meniere's disease; inner ear; endolymphatic sac drainage; steroids; declined surgery; natural course; Efficacy of steroids via endolymphatic sac; for intractable Meniere's disease
MeSH Terms: conditions — Meniere Disease | interventions — Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: endolymphatic sac drainage with steroids

SUMMARY:
Meniere's disease is a common inner ear disease with an incidence of 15-50 per 100,000 population. Since Meniere's disease is thought to be triggered by an immune insult to inner ear, we examined intra-endolymphatic sac application of large doses of steroids as de novo treatment for intractable Meniere's disease.

DETAILED DESCRIPTION:
Meniere's disease characterized by recurrent attacks of vertigo, fluctuating hearing loss and tinnitus, is a common disease with an incidence of 15-50 per 100,000 population. Some patients with Meniere's disease are strongly prevented from participating in activities of daily life and interaction with their social environment, such as work and schooling, due to frequent attacks of vertigo especially with progressive sensorineural hearing loss, in spite of various kinds of medication. This type of Meniere's disease is called intractable Meniere's disease. Although the oto-pathology in Meniere's temporal bones was revealed in 1938 to be inner ear endolymphatic hydrops, the definitive pathogenesis of Meniere's disease is still unknown and there is no radical treatment for this disease.

It has, however, been reported that Meniere's disease is usually triggered by immune, metabolic, infectious, traumatic or other insults to the inner ear, associated with a small misplaced malfunctioning endolymphatic sac. Among these insults, immune-mediated responses in the inner ear endo-organs such as the endolymphatic sac, stria vascularis and spiral ligament, are thought to be the main reason for the development of symptoms in Meniere's disease. Thus, systemic administration and/or local perfusion of corticosteroids into the middle ear have been adopted as an anti-immune or anti-inflammatory therapy for patients with intractable Meniere's disease. These treatments were reported to result in good relief from vertigo and improvement of hearing in some cases. However, these results especially for hearing did not last long enough to discontinue additional repetitive applications of steroids. Since Meniere's disease is characterized by repeated attacks of vertigo with fluctuating and/or progressive hearing loss unlike other inner ear diseases without recurrence such as sudden deafness and vestibular neuritis, it is necessary to refrain from repetitive applications of steroids for the long-term follow-up with Meniere's patients because of side effects.

For inner ear drug delivery, we noted another hopeful but unevaluated route, the longitudinal route from the endolymphatic sac to the cochlea and vestibule, suggested by several lines of evidence in animal studies. Morgenstern et al. and Lee et al. demonstrated that the intra-endolymphatic sac materials could reach the cochlear endolymphatic site through the vestibular aqueduct using a test marker and an oto-toxic drug, respectively. Recently, Yamasoba et al. suggested the possibility of gene therapy through the vestibular aqueduct route. We also revealed that intra-endolymphatic sac steroids could up-regulate a water channel molecule, aquaporin-3 mRNA in the cochlea.

In the present study, we examined the intra-endolymphatic sac application of large doses of steroids as de novo treatment for intractable Meniere's disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Meniere's Disease, who did not respond to various forms of medical and psychological managements for at least 6 months, i.e. intractable Meniere's disease.

Exclusion Criteria:

* Other known causes of vertigo including central lesion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 1996-04; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
the ratio of patients in vertigo supression and hearing improvement | post-operative 2-7 years

SECONDARY OUTCOMES:
the ratio of patients in canal improvement | post-operative 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tadashi Kitahara, M.D.,Ph.D., Principal Investigator — Department of Otolaryngology, Osaka University, School of Medicine
Locations (1):
- Department of Otolaryngology, Osaka University, School of Medicine, Suita, Osaka, Japan

REFERENCES:
- [Background] Kitahara T, Fukushima M, Uno Y, Mishiro Y, Kubo T. Up-regulation of cochlear aquaporin-3 mRNA expression after intra-endolymphatic sac application of dexamethasone. Neurol Res. 2003 Dec;25(8):865-70. doi: 10.1179/016164103771953989. PMID 14669532
- [Derived] Kitahara T, Horii A, Imai T, Ohta Y, Morihana T, Inohara H, Sakagami M. Effects of endolymphatic sac decompression surgery on vertigo and hearing in patients with bilateral Meniere's disease. Otol Neurotol. 2014 Dec;35(10):1852-7. doi: 10.1097/MAO.0000000000000469. PMID 24979126